CLINICAL TRIAL: NCT00994994
Title: Tranexamic Acid Reduces Blood Loss in Pediatric Cardiac Surgery
Brief Title: Tranexamic Acid in Pediatric Cardiac Surgery
Acronym: TXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okayama University (Other)
Responsible Party: Yuichiro Toda, Dept. of Anesthesiology, Okayama University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ped Txa Cya
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Blood Loss; Congenital Heart Disease
Keywords: pediatric cardiac surgery; bleeding; tranexamic acid; fibrinolysis; blood loss in pediatric cardiac surgery
MeSH Terms: conditions — Hemorrhage; Heart Defects, Congenital | interventions — Tranexamic Acid; Tranylcypromine; Antifibrinolytic Agents

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Active Comparator): 50 mg/kg of tranexamic acid was given as a bolus at the induction of anesthesia, followed by 15 mg/kg of continuous infusion and another 50 mg/kg into the bypass circuit.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): same volume of normal saline was given.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 50 mg/kg of tranexamic acid was given as a bolus at the induction of anesthesia, followed by 15 mg/kg of continuous infusion and another 50 mg/kg into the bypass circuit in TXA group. same volume of normal saline was given in Placebo group.
  Other Names: transamine; antifibrinolytic; lysin analogue

SUMMARY:
Tranexamic acid(TXA) is an antifibrinolytic agent to reduce blood loss in cardiac surgery. Previous seven RCTs comparing effects of TXA in pediatric cardiac surgery showed conflict results. The reason why they showed mixed results would be the imbalance of patients population with regard to presence of cyanosis. TXA would reduce blood loss in pediatric cardiac surgery with well balanced patients population.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* neonate born within 1 month
* preoperative inotropes
* preoperative mechanical ventilation
* preexisting coagulation disorder
* reoperation within 48 hours
* significant liver or kidney disease
* known allergy to TXA

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
the amount of blood loss (mediastinal and pericardial tube drainage) 24 hours after surgery | 24 hours after surgery

SECONDARY OUTCOMES:
blood loss 6 hours after surgery | 6 hours after surgery
the amount of blood transfusion | 24 hour after surgery
additional TXA administration | 24 hours after surgery
chest closure time (protamine to skin closure) | at the end of surgery
re-exploration of chest for excess bleeding | within 24 hours after surgery
duration of mechanical ventilation | at the time of extubation
length of stay in intensive care unit | at the time of discharge from ICU
episode of thrombotic complication | from drug administration to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yuichiro Toda, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Care, Okayama University Hospital

REFERENCES:
- [Derived] Shimizu K, Toda Y, Iwasaki T, Takeuchi M, Morimatsu H, Egi M, Suemori T, Suzuki S, Morita K, Sano S. Effect of tranexamic acid on blood loss in pediatric cardiac surgery: a randomized trial. J Anesth. 2011 Dec;25(6):823-30. doi: 10.1007/s00540-011-1235-z. Epub 2011 Sep 24. PMID 21947753